CLINICAL TRIAL: NCT05938049
Title: Carotid Doppler and Inferior Vena Cava Measuerments for Volume Guided Management in Acute Kidney Injury Patients
Brief Title: Carotid Doppler and IVC Measurements for Volume Guided Management in Acute Kidney Injury Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ayman Abdallah Mahmoud, principal investigator, Assiut University
Other Study IDs: CD&IVC in AKI
Record Dates: First submitted 2023-06-16; First posted 2023-07-10 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: patients whom fluid management will be guided by their IVC & carotid Doppler measurements
  Interventions: Device: IVC ultrasound & Carotid doppler
- Group B: patients in whom the fluid management will not guided by IVC & carotid Doppler measurements.

INTERVENTIONS:
Device: IVC ultrasound & Carotid doppler — bed side ultrasonographic assessement of inferior vena cava maximum and minimum diameters 2 to 5 cm caudal to its junction with the right atrium over a single respiratory cycle , inferior vena cava collapsibility index (IVC-CI) will calculated as (IVC max - IVC min)/IVC max).
  carotid doppler assessment (2-3 cm proximal to the carotid bulb in the longitudinal plane) of corrected carotid flow time(systole time/√cycle time) ,carotid artery peak velocity variation calculated as ([PV max- PV min]/PV mean) × 100, where PV mean = (PV max + PV min)/2. during three consecutive respiratory cycles. as part of their routine care and assessment
  Groups: Group A

SUMMARY:
1. Evaluate Inferior Vena Cava Indices (Diameters , IVC-CI)&carotid doppler measurements (corrected Carotid Flow Time ,Carotid Blood Flow ,Carotid Artery Peak Velocity Variations) as Non-Invasive Technique for volume guided management in AKI Patient.
2. Estimate correlation between IVC (Diameters , IVC-CI) & carotid doppler measurements (corrected Carotid Flow Time ,Carotid Blood Flow ,Carotid Artery Peak Velocity Variations) as Non-Invasive Technique for volume guided management in AKI Patient.

DETAILED DESCRIPTION:
Acute kidney injury affects increasing numbers of patients worldwide, it was estimated approximately 15% of all subjects treated in hospitals develop Acute kidney injury,even a small increase in serum creatinine may be associated with increased risk of mortality , Oliguric AKI it imposes a great challenge for fluid management.

Recently, ultrasonography for estimating volume status has been widely recommended because of its non-invasive nature, ease of acquisition, and reproducibility of measurements.Among these ultrasound modalities, ultrasonographic assessment of the inferior vena cava & Carotid doppler measurements .

In spontaneously breathing patients, the inferior vena cava (IVC) diameter and the IVC Collapsibility Index (IVC-CI) have been shown to correlate with the volume status and central venous pressure (CVP) . also has been shown to indicate fluid status in children , ventilated patients and healthy volunteers .

corrected Carotid Flow Time (CFT) unaffected by respiration predicting fluid responsiveness that has shown promising results.Studies to date have shown that corrected CFT increases in response to fluid administration or consumption , and decreases in response to volume removal in dialysis and blood donation .

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with Acute Kidney Injury
2. age must be more than 18 years

Exclusion Criteria:

1. Morbid obesity (BMI >35)
2. End Stage Renal Disease (ESRD) on dialysis
3. Sever ventricular dysfunction, valvular heart disease
4. Carotid stenosis >50%
5. chronic obstructive pulmonary disease.
6. Pregnancy & tense ascites

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: consecutive Patients admitted to hospital with AKI or developing AKI during hospital admission course (AKI can be defined according to the Kidney Disease: Improving Global Outcomes (KDIGO) guidelines either an elevation in serum creatinine (≥ 26.5 µmol/L or ≥1.5 folds of base line) or a reduced urine output (<0.5 ml/kg/h for 6 hours or more))
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
percentage of participants with improved serum creatinine level in µmol/L in groups A and B. | at 48 hours
  percentage of participants with improved serum creatinine level in µmol/L in groups A and B.
percentage of participants with improved urine out put in ml/kg/h in groups A and B. | at 48 hours
  percentage of participants with improved urine out put in ml/kg/h in groups A and B.

SECONDARY OUTCOMES:
percentage of participants with improved mean arterial blood pressure in mmHg in groups A and B. | at 48 hours
  percentage of participants with improved mean arterial blood pressure in mmHg in groups A and B.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Saxena A, Meshram SV. Predictors of Mortality in Acute Kidney Injury Patients Admitted to Medicine Intensive Care Unit in a Rural Tertiary Care Hospital. Indian J Crit Care Med. 2018 Apr;22(4):231-237. doi: 10.4103/ijccm.IJCCM_462_17. PMID 29743761
- [Background] Miller TE, Bunke M, Nisbet P, Brudney CS. Fluid resuscitation practice patterns in intensive care units of the USA: a cross-sectional survey of critical care physicians. Perioper Med (Lond). 2016 Jun 16;5:15. doi: 10.1186/s13741-016-0035-2. eCollection 2016. PMID 27313844
- [Background] Thanakitcharu P, Charoenwut M, Siriwiwatanakul N. Inferior vena cava diameter and collapsibility index: a practical non-invasive evaluation of intravascular fluid volume in critically-ill patients. J Med Assoc Thai. 2013 Mar;96 Suppl 3:S14-22. PMID 23682518
- [Background] Levine AC, Shah SP, Umulisa I, Munyaneza RB, Dushimiyimana JM, Stegmann K, Musavuli J, Ngabitsinze P, Stulac S, Epino HM, Noble VE. Ultrasound assessment of severe dehydration in children with diarrhea and vomiting. Acad Emerg Med. 2010 Oct;17(10):1035-41. doi: 10.1111/j.1553-2712.2010.00830.x. PMID 21040103
- [Background] Barbier C, Loubieres Y, Schmit C, Hayon J, Ricome JL, Jardin F, Vieillard-Baron A. Respiratory changes in inferior vena cava diameter are helpful in predicting fluid responsiveness in ventilated septic patients. Intensive Care Med. 2004 Sep;30(9):1740-6. doi: 10.1007/s00134-004-2259-8. Epub 2004 Mar 18. PMID 15034650
- [Background] Blehar DJ, Glazier S, Gaspari RJ. Correlation of corrected flow time in the carotid artery with changes in intravascular volume status. J Crit Care. 2014 Aug;29(4):486-8. doi: 10.1016/j.jcrc.2014.03.025. Epub 2014 Apr 2. PMID 24930363
- [Background] Hossein-Nejad H, Mohammadinejad P, Lessan-Pezeshki M, Davarani SS, Banaie M. Carotid artery corrected flow time measurement via bedside ultrasonography in monitoring volume status. J Crit Care. 2015 Dec;30(6):1199-203. doi: 10.1016/j.jcrc.2015.08.014. Epub 2015 Aug 22. PMID 26410681
- [Background] Doctor M, Siadecki SD, Cooper D Jr, Rose G, Drake AB, Ku M, Suprun M, Saul T. Reliability, Laterality and the Effect of Respiration on the Measured Corrected Flow Time of the Carotid Arteries. J Emerg Med. 2017 Jul;53(1):91-97. doi: 10.1016/j.jemermed.2017.01.056. Epub 2017 Mar 25. PMID 28351511
- [Background] Shokoohi H, Berry GW, Shahkolahi M, King J, King J, Salimian M, Poshtmashad A, Pourmand A. The diagnostic utility of sonographic carotid flow time in determining volume responsiveness. J Crit Care. 2017 Apr;38:231-235. doi: 10.1016/j.jcrc.2016.10.025. Epub 2016 Nov 9. PMID 27987483
- [Background] Mackenzie DC, Khan NA, Blehar D, Glazier S, Chang Y, Stowell CP, Noble VE, Liteplo AS. Carotid Flow Time Changes With Volume Status in Acute Blood Loss. Ann Emerg Med. 2015 Sep;66(3):277-282.e1. doi: 10.1016/j.annemergmed.2015.04.014. Epub 2015 May 21. PMID 26003002